CLINICAL TRIAL: NCT06045052
Title: An Open-label, Phase II Study to Assess the Efficacy and Safety of Eltrombopag for the Treatment of Children and Adolescents With Fanconi Anemia.
Brief Title: Eltrombopag for Treatment of Fanconi Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Julian Sevilla (Other)
Responsible Party: Sponsor-Investigator, Julian Sevilla, Dr. Julián Sevilla Navarro, MD, PhD, Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Organization: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FANCREV
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag will be administered orally once daily for 24 weeks (6 months) and the dose will be adjusted according to race, age and weight. Patients who achieve at least partial remission may continue treatment for up to one year.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag tablets by mouth once daily for 24 weeks (6 months) with the dose depending on race, age and weight.
  Other Names: Revolade®

SUMMARY:
An open-label, phase II study to assess the efficacy and safety of eltrombopag for the treatment of children and adolescents with Fanconi anemia.

DETAILED DESCRIPTION:
Open-label, phase II study to assess the efficacy and safety of eltrombopag in the treatment of patients diagnosed with Fanconi anemia who have no immediate curative treatment for their bone marrow failure (n=10). The primary objective of this open-label, phase II proof of concept study is to assess the efficacy and safety of using eltrombopag for the treatment of patients with FA before conducting a larger phase II/III study.

Specific objectives:

* Primary: To assess the efficacy of eltrombopag on hematopoiesis by measuring changes in peripheral platelet, hemoglobin and neutrophil counts.
* Secondary: To assess the safety of eltrombopag in patients with Fanconi anemia. If the preliminary efficacy and safety results from the study are positive, we will propose its expansion to a multi-institutional Phase II/III study within the framework of the Spanish Fanconi Anemia Research Network.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Fanconi anemia. Diagnosis will be defined by the presence of biallelic mutations in genes known to cause the disease and/or by positive chromosome breakage analysis of lymphocytes and/or skin fibroblasts (for cases of mosaicism).
* Age from 4 to ≤ 17 years.
* Lansky index > 80%.
* Informed consent provided in accordance with current legislation.
* Presenting with one or more of one of the following clinically significant cytopenias:

platelet count ≤ 50x109/L or transfusion dependence, having required at least 2 transfusions in the 8 weeks prior to inclusion in the study; granulocyte count < 0.75x109/L; hemoglobin < 9 gr/dL or transfusion-dependent anemia having received 2 transfusions in the 8 weeks prior to inclusion in the study.

Exclusion Criteria:

* Patients with HLA-matched related donor or unrelated donor with a 12/12 match who is immediately available.
* Evidence of myelodysplastic syndrome or leukemia or cytogenetic abnormalities predictive of these disorders in bone marrow aspirates. In the event, the evaluations performed two months before patient inclusion in the clinical study will be considered valid.
* Baseline creatinine greater than 2.5 times the upper limit of normality.
* GOT/AST or GPT/ALT more than three times the upper limit of normality. Direct bilirubin greater than 1.5 times the upper limit of normality.
* Patients who are already receiving treatment with some drug for bone marrow failure may be included as long as the dose administered remains stable for at least two months. In the event that such treatment requires an increase in dose during the study, the patient must withdraw from the trial. Patients who have already started Revolade® treatment in the previous two months may also be included, and the blood counts and baseline bone marrow studies performed at the start of treatment will be used.
* Women of postpubertal age and therefore at risk of pregnancy should have a negative serum or urine pregnancy test at the screening visit and agree to use a contraceptive method throughout the treatment period and for at least one month after.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Assessing the efficacy of eltrombopag on hematopoiesis | 6 months
  An analysis of the proportion of patients with complete response and/or partial response after 6 months of treatment in the absence of transfusions or rescue therapy will be performed.

SECONDARY OUTCOMES:
Evaluation of the incidence of clonal evolution | 6 and 12 months.
  Monitoring of cytogenetic abnormalities or specific mutations related to hematologic malignancies at months 6 and 12 from start of treatment.
Identification and tracking of adverse reactions associated with eltrombopag treatment in patients with Fanconi anemia graded | 3, 6, 9 ans 12 months.
  The CTCAE version 5.0 criteria will be used at 3, 6, 9 and 12 months from start of treatment.
Determination of the proportion of grafted cells | 12 months
  It will be evaluated in patients seen to have reverted cells, involving either correction of a pathogenic mutation (natural mosaicism) or due to the infusion of hematopoietic stem cells transduced with the lentiviral vector carrying the FANCA gene

CONTACTS AND LOCATIONS:
Overall Officials: Julián Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús (HIUNJ)
Locations (1):
- Hospital Infantil Universitario Niño Jesús (HIUNJ), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Iriondo J, Zubicaray J, Rio P, Catala A, Solsona M, Sanz A, Gomez A, Sebastian E, de la Cruz A, Galan A, Navarro S, Larcher L, de Andoin NG, Uriz JJ, Vagace JM, Gonzalez de Pablo J, Pujol MR, Nicoletti E, Surralles J, Martin-Prado S, Schwartz JD, Soulier J, Bueren JA, Sevilla J. Eltrombopag for Bone Marrow Failure in Fanconi Anemia: Results From the Phase II Clinical Trial FANCREV. Eur J Haematol. 2025 Oct;115(4):403-412. doi: 10.1111/ejh.70007. Epub 2025 Jul 16. PMID 40665878